CLINICAL TRIAL: NCT05289375
Title: Efficacy of the Vacucis Candida® Autovaccine in the Management of Chronic Oral Candidiasis. Randomized Triple-blind Randomized Clinical Trial.
Brief Title: Efficacy of the Vacucis Candida® Autovaccine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Mario Pérez Sayáns, Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RCT-VCA-22
Record Dates: First submitted 2022-02-11; First posted 2022-03-21 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Oral Candidiasis; Oral Candidiasis Recurrent; Radiotherapy; Complications; Candida Albicans Infection; Microbial Colonization; Xerostomia
Keywords: oral candidiasis
MeSH Terms: conditions — Candidiasis, Oral; Communicable Diseases; Xerostomia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (T) (Active Comparator): Group formed by those patients who will receive the drug to be tested Vacucis
  Interventions: Drug: Vacucis autovaccine
- Placebo control group (P) (Placebo Comparator): Group formed by those patients who will receive placebo, in the same dosage and duration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vacucis autovaccine — A sample will be taken from all participants in group T following the manufacturer's instructions for the design of the autovaccine, using a sterile swab that will be placed in a transport medium and sent to the laboratory. After 1 month from the sample collection, the laboratory will send in a container/dispenser (with the same appearance in both groups) to the T group will be administered the complete autovaccine ((with two applications per day for 7 weeks)
  Arms: Test group (T)
Drug: Placebo — A sample will be taken from all participants in group P following the manufacturer's instructions for the design of the autovaccine, using a sterile swab that will be placed in a transport medium and sent to the laboratory (as in group T). After 1 month from the collection of the sample, the laboratory will send it in a container/dispenser (with the same appearance in both groups). The content in group P will receive a placebo in the same dosage and temporality as group T, it will be the same except for the active ingredient, that is, only thimerosal, methylcellulose, sodium chloride and orange essence.
  Arms: Placebo control group (P)

SUMMARY:
Introduction: Oral candidiasis is an infectious disease caused by the growth of Candida colonies and their penetration into oral tissues when physical barriers and host defenses are weakened. It constitutes one of the most common pathologies within the field covered by Dentistry. Candida infections are found in at least 80% of AIDS patients and in a third of HIV infection cases. Systemic diseases such as diabetes and a wide pharmacological arsenal to which the general population is subjected, are other causes of the increase in the prevalence of this disease. In addition, the high prevalence of oral sequelae (hyposialia) in the population over 65 years of age, due to the specific characteristics of this age group, such as multiple pathologies and drug use, explains the presence of this disease in this segment. of the population One of the great difficulties for the study of this disease is the diversity of predisposing factors, which do nothing but throw greater confusion into the results of the different works.

Objective: To evaluate the reduction/suppression of signs and symptoms of oral candidiasis in patients treated with head and neck RT, users of Vacucis or Placebo.

Material and method: Patients will receive information regarding the trial and, if they meet the inclusion criteria and agree to participate in it, they will sign the informed consent. All patients will be informed following the usual care practice of the characteristics of their candidiasis infection as well as the possibilities and alternatives of treatment and their respective efficacy.

A descriptive analysis of the sample in terms of prevalence will be carried out. Categorical variables will be described as frequency and percentage and continuous variables as mean and standard deviation or median and interquartile range depending on their adjustment to normality, which will be calculated with the Kolmogorov-Smirnov test. To study the effect of the vaccine on the evolution of candidiasis, the Chi-square test, Student's t test or the non-parametric Mann-Whitney test will be used. The association of prevalence with CFU in both groups will be analyzed using the ANOVA test. Those values of p < 0.05 will be considered significant.

DETAILED DESCRIPTION:
The design of a randomized, randomized (test and placebo) triple-blind (patient, investigator and evaluator) clinical trial is proposed. The clinical trial will be carried out in accordance with the criteria recommended in the CONSORT Guidelines.

All patients who agree to participate will have a sample taken following the manufacturer's instructions for the design of the autovaccine, using a sterile swab that will be placed in transport medium (AMIES type) and sent to the laboratory. After 1 month of taking the sample, the laboratory that will be in possession of the randomization will damage the container/dispenser, which will be exactly the same in both groups T and P. Group T will be administered the complete autovaccine, while group P , the content will be the same except for the active ingredient, that is, only thimerosal, methylcellulose, sodium chloride and orange essence. In this way, neither the research group nor the patient himself will be known by the group to which he has been assigned.

In the event of unforeseen adverse effects, which are not expected, patients will be withdrawn from the study and treated according to standard care practice. All patients will be able to resort to rescue medication if the symptomatology is exacerbated during the follow-up period of the study, always under the prescription of the physician (nystatin aqueous rinse solution 1ml/100,000 IU or oral Fluconazole 50 mg/24 hours).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of RT in the head and neck region that directly or indirectly involves any of the jaws.
* Adult patients
* Hemodynamically stable patients without contraindications to receive an autovaccine (see exclusion)
* Patients with a stable oncological situation without active tumor
* Patients who present candidiasis demonstrated by clinical examination (signs and symptoms of candidiasis) and microbiological (culture).

Exclusion Criteria:

* Minor patients
* Pregnant patients
* Patients with an unstable medical situation, both from a hemodynamic and oncological point of view (advanced tumors with metastases, recurrences or inoperable tumors)
* Patients undergoing treatment with CT that involves an affectation of the immune system
* Patient under treatment with antifungals for mycoses of any origin
* Allergy to the active substance or to any of the other components of Vacucis.
* Serious disorders of the immune system.
* Diseases that severely affect immunity.
* Presence of fever.
* People with allergies to yeasts
* People with allergy to chloramphenicol
* Patients treated with MAOIs (monoamine oxidase inhibitors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms of candidiasis | 6 months
  Mouth pain will be measured with the visual analog scale. It consists of a 10cm straight line with the words "No Pain" on the left end and "Worst Pain Imaginable" on the right end. Minimum value 0, maximum value 10. A value lower than 4 on the VAS means mild or mild-moderate pain, a value between 4 and 6 implies the presence of moderate-severe pain, and a value higher than 6 implies the presence of very severe pain.
Oral signs of candidiasis | 6 months
  Prosthetic stomatitis will be evaluated according to Newton's clinical classification. Grade I: Reddish stippling. Grade II: Diffuse erythema. Grade III: Granular mucosa and non-neoplastic papillary hyperplasia.
Modification of fungal growth | 6 months
  It will be evaluated with the microbiological study: the CFU (or colony forming units) will be studied in culture plates.
Determination of quality of life | 6 months
  It will be assessed with the oral health impact profile (OHIP-14). This questionnaire includes seven dimensions with 14 items to determine the quality of life. The higher the average value of the seven dimensions, the more negative the impact of oral health on the quality of life of an individual.Minimum of 0 points and maximum of 56 points.

SECONDARY OUTCOMES:
Relationship between clinical signs and symptoms and saliva levels. | 6 months
  The patient's saliva will be quantified by salivometry using: TSG-I: basal global saliva rate and TSG-II: stimulated global saliva rate.
Relationship between clinical signs and symptoms and xerostomia | 6 months
  The degree of xerostomia (subjective sensation) will be evaluated through the xerostomia inventory test (XI).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We will anonymize and categorize the clinical data of the patients to share the information with the other researchers of the group.